CLINICAL TRIAL: NCT03192748
Title: A Registry Study of Runzaozhiyang Capsule Used in Clinical Real World
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Yanming Xie, Deputy director, China Academy of Chinese Medical Sciences
Other Study IDs: Runzao
Record Dates: First submitted 2017-06-14; First posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Eczema
MeSH Terms: conditions — Eczema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is get to know what and how Runzaozhiyang capsule in hospital results in drug-induced liver injury or adverse drug reactions from a cohort event monitoring as registration research.

DETAILED DESCRIPTION:
In order to improving monitoring drug-induced liver injury or adverse drug reactions of Chinese medicine containing Radix Polygoni Multiflori in clinical real world, registry study is suitable method in this area. Otherwise, nested case control study is used to find out the mechanism of drug-induced liver injury. Calculate the incidence of drug-induced liver injury or adverse drug reactions is one of the main aims for this study. Safety surveillance on Chinese medicine containing Radix Polygoni Multiflori is an important problem that needs to be sorted out through large sample observational study. According to the relevant regulations of the CFDA, 3000 cases need to be registered at least. The aim population is who using Runzaozhiyang capsule 's with abnormal liver function before medication from June 2017 to June 2019.

ELIGIBILITY:
Inclusion Criteria:

Patients using Runzaozhiyang capsule 's with abnormal liver function before medication from June 2017 to June 2019.

Exclusion Criteria:

none

Min Age: 1 Hour | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The aim population for observation is who using Runzaozhiyang capsule 's with abnormal liver function before medication from June 2017 to June 2019.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-06-19 (Estimated); Primary Completion 2017-06-19 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Is there any abnormality in liver function test index（ALT、AST、TBil、GGT） after using runzaozhiyang capsule around two weeks later? | After using runzaozhiyang capsule around two weeks later.
  Based on data from the National Center for adverse drug reactions (ADR), Chinese herbal medicine containing Polygonum multiflorum may cause liver damage, but further confirmation is needed.The liver function includes glutamic-pyruvic transaminase,glutamic-oxalacetic transaminase,GGT,TBil.

SECONDARY OUTCOMES:
Is there any abnormality in renal function test index（Bun、Cr） after medication? | After using runzaozhiyang capsule around two weeks later.
  Observation of whether the kidney function damage after treatment.The renal function includes creatinine,usea nitrogen.
Is there any abnormality in ECG after medication? | After using runzaozhiyang capsule around two weeks later.
  Observation of whether the ECG damage after treatment.ECG is the most common method of detection of myocardial ischemia and the diagnosis of angina pectoris.
Is there any abnormality in basic life sign（body temperature, blood pressure and pulse）？ | During using runzaozhiyang capsule around two weeks.
  Observation of whether the basic life sign damage after treatment.In the medical care system, body temperature, blood pressure and pulse are the most important and basic three physiological parameters of the vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Yanming Xie, BA, Principal Investigator — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences

IPD SHARING:
Plan to Share IPD: No